CLINICAL TRIAL: NCT03055598
Title: Effect of Auryxia on ESA Utilization in ESRD Patients With High Ferritin & Low Transferrin Saturation: A Pilot Project
Brief Title: Ferric Citrate in ESRD Pilot Project
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sreedhar Mandayam (Other)
Collaborators: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Sreedhar Mandayam, MD, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-39364 Ferric Citrate in ESRD
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: End Stage Renal Disease; Chronic Kidney Diseases
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — ferric citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferric Citrate (Experimental): Ferric Citrate (Auryxia) will be dosed initially at 2 tablets three times a day (with meals).
  Interventions: Drug: Ferric Citrate

INTERVENTIONS:
Drug: Ferric Citrate — Doses can be adjusted as needed by 1 to 2 tablets up to a maximum of 12 tablets daily. Dose can be titrated at 1-week or longer intervals.
  Other Names: Auryxia

SUMMARY:
This research study is for participants that have End Stage Renal Disease (ESRD). ESRD is the last stage of chronic kidney disease. Anemia is very common in ESRD patients and require erythropoiesis-stimulating agents (ESAs) for treatment. Anemia happens when there are not enough red blood cells in your body. ESAs work by helping the bone marrow to produce red blood cells. There are two ESAs licensed for the treatment of anemia of Chronic Kidney Disease (CKD) in the Unites States: epoetin alfa and darbopoetin alfa. ESA therapy is considered safe. However, major adverse effects should be acknowledged, including an increased risk of death, thromboembolic complications, stroke, heart attack, aplastic anemia, tumor progression, and others. To minimize risks of these adverse events, careful monitoring of hemoglobin levels, along with adjustment of ESA dosing, to maintain the lowest hemoglobin level clinically needed is recommended.

Ferric Citrate, also called Auryxia, is an iron-based phosphate binder that may decrease ESA usage while maintaining hemoglobin levels. Phosphate binders are medications used to reduce the body's absorption of phosphate. In a prior study, it was seen that some laboratory values, such as iron levels, changed positively in response to Auryxia. In this study we want to see if using Auryxia will cause a change in laboratory values and lower the use of ESAs in ESRD patients.

DETAILED DESCRIPTION:
Iron deficiency anemia is very prevalent in end stage renal disease (ESRD) patients. Patients with ESRD require phosphate binders for hyperphosphatemia and erythropoiesis-stimulating agents (ESAs) and intravenous (IV) iron for anemia. In patients with ESRD, iron deficiency occurs more frequently, because of increased external losses of iron, decreased availability of the body's storage of iron, and perhaps a deficit in intestinal iron absorption.

ESRD patients tend to lose about 3 grams of iron every year from chronic bleeding, frequent phlebotomy and blood trapping in the dialysis apparatus. Total body iron stores of about 20-25 mg are mostly maintained by recycling from senescent red blood cell (RBC) count by macrophages of the reticulo-endothelial system. In addition, to true iron deficiency, many ESRD patients have functional iron deficiency, characterized by impaired iron release from body stores that is unable to meet the demand for erythropoiesis (also called reticuloendothelial cell iron blockade). These patients have low serum transferrin saturation (TSAT, a measure of circulating iron) and normal or high serum ferritin (a marker of body iron stores). Dietary iron absorption under usual circumstances accounts for only 1-2 mg/day and is almost equal to daily iron losses from intestinal and skin cell shedding.

For treatment of anemia caused by chronic renal disease, the United States Food and Drug Administration (FDA) has approved the use of ESA therapy. There are two ESAs licensed for the treatment of anemia of CKD in the Unites States: epoetin alfa and darbopoetin alfa. Both are glycoproteins that are manufactured using recombinant DNA technology. They stimulate erythropoiesis through the same mechanism of action as endogenous erythropoietin. The starting dose of epoetin is 50 units/kg (3000-4000 units/dose) once or twice a week, and darbepoetin is started at 0.45 mcg/kg and can be administered every 2-4 weeks. To avoid impaired erythropoiesis caused by true iron deficiency or functional iron deficiency, iron stores should be fully replenished before and during ESA therapy. ESA therapy is considered safe. However, major adverse effects should be acknowledged, including an increased risk of death, thromboembolic complications, stroke, heart attack, aplastic anemia, tumor progression, and others. To minimize risks of these adverse events, careful monitoring of hemoglobin levels, along with adjustment of ESA dosing, to maintain the lowest hemoglobin level clinically needed is recommended.

Given that ESRD is a pro-inflammatory condition, substantial elevation in serum ferritin is very common in ESRD patients. The role of iron replacement therapy in ESRD patients with high serum ferritin but low transferrin saturation is not clear at all. In fact, most anemia management protocols recommend stopping iron replacement when ferritin levels are greater than 1,200 ng/ml, even if the TSAT is below 20%. The United States Renal Data System (USRDS) reports for that 55% of prevalent ESRD patients (2012-2014) have a ferritin >800 ng/ml and 22% had ferritin>1200 ng/ml. In one of our local dialysis centers, close to 45% of patients seem to have a ferritin greater than 1,200 ng/ml and about 20% have a combination of low TSAT and high ferritin.

Ferric citrate (Auryxia) is a novel, iron-based phosphate binder that increases iron stores and decreases IV iron and ESA usage while maintaining hemoglobin levels, and may decrease the cost of ESRD care. By binding phosphate in the GI tract and decreasing absorption, ferric citrate lowers the phosphate concentration in the serum. In addition to effects on serum phosphorus levels, Auryxia has been shown to increase serum iron parameters, including ferritin, iron and TSAT. In dialysis patients treated with Auryxia in a 52-week study in which IV iron could also be administered, mean (SD) ferritin levels rose from 593 (293) ng/mL to 895 (482) ng/mL, mean (SD) TSAT levels rose from 31% (11) to 39% (17) and mean (SD) iron levels rose from 73 (29) mcg/dL to 88 (42) mcg/dL. In contrast, in patients treated with active control, these parameters remained relatively constant.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study specific procedures
2. Male and females aged 18 years and older
3. In the Investigator's opinion, expected to survive at least 3 months
4. Able to tolerate phosphate binders
5. ESRD and on dialysis for over 90 days
6. Deemed stable by Investigator
7. Serum Ferritin >1000 ng/ml (measured as average of at least 2 values in the last 3 months +/- 10 days)
8. TSAT < 30% ( measured as average of at least 2 values in the last 30 days, +/- 10 days)
9. Hemoglobin < 12g/dl (measured as average of at least 2 values in the last 30 days, +/- 10 days)
10. Currently on ESA for at least 1 month, as per dialysis unit protocol

Exclusion Criteria:

1. Inability or refusal to give informed consent
2. Subject unwilling to take study medication for 3 months
3. Currently on IV Iron
4. Currently on Auryxia as phosphate binder (or received in prior 3 months)
5. Deemed non-compliant by care team for dialysis or medication
6. Active gastrointestinal bleed
7. Inflammatory bowel disease
8. History of malignancy within 5 years before screening (exceptions: squamous and basal cell carcinomas of the skin and carcinoma of the cervix in situ, or a malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence).
9. Known allergy to oral iron products
10. Pregnant
11. Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
change in average weekly ESA dose determination from baseline to day 90 | day 90
  determine change in average dose of ESA use when using Auryxia
change in mean serum iron from baseline to day 90 | day 90
  assess change in mean serum iron while using Auryxia
change in mean ferritin from baseline to day 90 | day 90
  assess change in mean ferritin while using Auryxia

SECONDARY OUTCOMES:
change in average weekly ESA dose determination | baseline, day 30, day 60
  determine change in average dose of ESA use when using Auryxia
change in mean serum iron | baseline, day 30, day 60
  assess change in mean serum iron while using Auryxia
change in mean ferritin | baseline, day 30, day 60
  assess change in mean ferritin while using Auryxia
TSAT value | baseline, day 30, day 60, day 90
  values if less than 30% to greater than 30% to determine effectiveness
hemoglobin value | baseline, day 30, day 60, day 90
  elevated serum ferritin (>1000 ng/ml) to determine effectiveness
Kidney Disease Quality of Life (KDQOL)-36 energy score | Baseline and 90 days
  KDQOL-36 energy score to determine overall quality of life
KDQOL-36 fatigue score | Baseline and 90 days
  KDQOL-36 fatigue score to determine overall quality of life
KDQOL-36 depression score | Baseline and 90 days
  KDQOL-36 depression score to determine overall quality of life
Number of participants alive or dead (Survival status) at 90 days | at 90 days
  Measured by death (yes/no) and date

CONTACTS AND LOCATIONS:
Overall Officials: Sreedhar Mandayam, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Harris Health System - Riverside Dialysis Center, Houston, Texas
  - US Renal Care- Scott Street, Houston, Texas

IPD SHARING:
Plan to Share IPD: No